CLINICAL TRIAL: NCT00178464
Title: Aspirin Prophylaxis in Sickle Cell Disease
Acronym: START
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: University of Miami (Other); Bayer (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09661; 5R01NS045948-03 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2012-01-04 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; hemoglobin SS disease; hemoglobin S Beta-0 Thalassemia; silent infarction in sickle cell disease; overt stroke in sickle cell disease; aspirin; transcranial Doppler ultrasound; neurocognitive testing
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aspirin (Experimental): One-arm study
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: aspirin — 81 mg flavored chewable tablets. Subjects between the ages of 2.0 and 4.99 years will receive half of an 81 mg aspirin tablet each day. Those older than 5.0 years will receive a daily 81 mg aspirin tablet. The subject will receive the study drug for a period of 12 months.
  Other Names: Acetylsalicyclic Acid; ASA

SUMMARY:
Neurologic complications secondary to cerebrovascular damage are prevalent in children with sickle cell disease. These patients experience both clinically overt cerebrovascular accidents and "silent infarctions" demonstrated by magnetic resonance imaging (MRI). They are also at risk for neurocognitive abnormalities.We hypothesize that daily, low-dose aspirin therapy will safely diminish the incidence and progression of cognitive deficits as well as the predisposition to overt and silent stroke in children with homozygous sickle cell disease (Hgb SS) or hemoglobin S Beta Zero Thalassemia (Hgb SB-0 Thal). In order to optimize the design of a future trial to test this hypothesis, we propose a pilot study to test the safety and tolerability of aspirin in young children with sickle cell disease.

DETAILED DESCRIPTION:
The trial's primary objective is to evaluate the safety and tolerability of daily low-dose aspirin in children with sickle cell disease. The secondary objectives are to assess (1) The feasibility of recruiting children with Hgb SS and Hgb S Beta-0 Thalassemia to an aspirin trial, (2) The level of compliance with aspirin administration in the proposed patient population, (3) The most useful assessments in a battery of age-appropriate neurocognitive tests, (4) The feasibility of magnetic resonance imaging (MRI) and magnetic resonance angiography (MRA) studies and the utility of classification systems for use in group comparisons, (5) Preliminary data regarding trends in transcranial Doppler (TCD) ultrasound velocities over time and the validity of using trends for group comparisons, (6) Preliminary data regarding the effect of aspirin therapy on the incidence of cognitive deficit, imaging changes, overt stroke, painful crises, and acute chest syndrome. Subjects will include children between the ages of 2 and 7.99 years with documented Hgb SS or Hgb S Beta-0 Thalassemia who are followed at Golisano Children's Hospital at Strong and the University of Miami. All subjects will receive daily aspirin (about 2.5 - 5.1 mg/kg daily). Subjects will receive therapy for 12 months. There will be careful laboratory and clinical monitoring every 3-6 months and more frequently if needed. Pre and post treatment clinical complications, neurocognitive testing, MRI, MRA, and TCD studies will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Children ages 2 - 7.99 years with a diagnosis of Hb SS or Hb Sß0 thalassemia, documented by hemoglobin electrophoresis and a complete blood count (CBC). 2. Influenza vaccination during the previous year or intended before the upcoming flu season. 3. Evidence of past infection with, or immunization against, varicella. 4. Negative pregnancy tests in girls of childbearing potential. 5. Informed consent signed by the parent or legal guardian.

Exclusion Criteria:

* 1. Prior history of overt stroke or cerebral hemorrhage. 2. Known history of allergic reaction to aspirin. 3. History of Reye's syndrome 4. Diagnosis of G-6-PD deficiency or von Willebrand's disease 5. Prolongation of the bleeding time or abnormal closure time, prothrombin time (PT), or partial thromboplastin time (PTT). 6. Active gastrointestinal (GI) bleeding or a history of GI bleeding. 7. Hepatic disease (AST or ALT >2x upper limit of normal, Direct bilirubin > 1.5 mg/dL) or renal disease (creatinine >2x upper limit of normal or 2 mg/dl, whichever is smaller). The exclusion criteria laboratory study ranges have been specified as greater than 2 times the upper limit of normal. 8. Hypertension (BP >95% for age and height). 9. Current treatment with chronic transfusion therapy. 10. Evidence of hemorrhage on MRI. 11. A mean TCD velocity > 200 cm/sec. in the middle cerebral artery (MCA) or internal carotid artery (ICA). 12. Evidence of Moyamoya syndrome on MRA. 13. Evidence of pregnancy. 14. Evidence of an inability to comply with testing procedures. 15. Inability to provide informed consent.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2005-03; Primary Completion 2009-04 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norma B. Lerner, MD, Principal Investigator — University of Rochester

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin: Aspirin 81 mg flavored chewable tablets. Subjects between the ages of 2.0 and 4.99 years will receive half of an 81 mg aspirin tablet each day. Those older than 5.0 years will receive a daily 81 mg aspirin tablet. The subject will receive the study drug for a period of 12 months.
Period: Overall Study
Arm/Group | Aspirin
Started | 11
Completed | 9
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aspirin
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events
Description: Occurrence of individual serious adverse events and relationship to aspirin
Time Frame: 12 months
Population: Intention to treat
Measure: Number; unit: events
Arm/Group | Aspirin
Number analyzed (Participants) | 8
events
  No relationship | 6
  Unlikely | 9
  Possible | 0
  Probable | 0
  Definite | 0

2. Secondary Outcome: # of Subjects Recruited Over Time, Screening Failures, Withdrawal Rates;Compliance (Pill Counts & Labs);Changes in Performance on Neurocognitive Tests; Changes in MRI/MRA; Changes in TCD;Incidences of Stroke, Acute Chest Crises, and Pain Crises
Time Frame: 12 months
Reporting Status: Not Posted

3. Primary Outcome: Number of Adverse Events
Description: Occurrence of individual adverse events and relationship to aspirin
Time Frame: 12 months
Population: Intention to treat
Measure: Number; unit: events
Arm/Group | Aspirin
Number analyzed (Participants) | 8
events
  No relationship | 8
  Unlikely | 3
  Possible | 5
  Probable | 1
  Definite | 2

ADVERSE EVENTS:
Arm/Group | Aspirin
Serious Adverse Events (participants affected / at risk) | 8/11
Other Adverse Events (participants affected / at risk) | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=11)
Fever resulting in Hospitalization (General disorders) | 6 (7) — may be in association w/another SAE
Severe Anemia resulting in hospitalization (Blood and lymphatic system disorders) | 1 (1) — may be assoc w/other SAEs.
Pneumonia resulting in hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vasoocclusive Crisis Pain resulting in hospitalization (Musculoskeletal and connective tissue disorders) | 2 (6) — May be assoc w/other SAEs.
Splenic Sequestration (Blood and lymphatic system disorders) | 1 (1) — May be associated w/other SAEs.
Asthma resulting in hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) — May be assoc w/other SAEs.
Fracture resulting in hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute Chest Syndrome resulting in hospitalization. (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abnormal MRA resulting in withdrawal from study. (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=11)
Fever (General disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scabies (Skin and subcutaneous tissue disorders) | 1 (1)
Bleeding per rectum (Blood and lymphatic system disorders) | 1 (3)
Epistaxis (Blood and lymphatic system disorders) | 2 (3)
Pain (General disorders) | 3 (3)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (1)
Otitis Media (Ear and labyrinth disorders) | 1 (1)
Allergic reaction (General disorders) | 1 (1)
Tarry stool (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No